CLINICAL TRIAL: NCT06182527
Title: Evaluation of the Everyday Relevance of Reactive Hypoglycemia in the Oral Glucose Tolerance Test Using Continuous Glucose Measurement.
Brief Title: Relevance of Reactive Hypoglycemia During an OGTT in Everyday Life Using Continuous Glucose Measurement
Acronym: HypoCGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Prof. Martin Heni, University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 147/2023
Record Dates: First submitted 2023-11-27; First posted 2023-12-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hypoglycemia, Reactive
Keywords: Reactive Hypoglycemia; Oral glucose tolerance test; Continuous glucose monitoring
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Masking Description: Every participant receives a Freestyle Libre PRO IQ Sensor, a system which ensures blinding of the glucose levels to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM Group (Experimental): Every participant receives a Free Style Libre Pro IQ sensor for 14 days. Glucose levels will be recorded. In addition perception of hypoglycemia and counter action will be assessed.
  Interventions: Device: Free Style Libre Pro IQ

INTERVENTIONS:
Device: Free Style Libre Pro IQ — Every participant receives a Free Style Libre Pro IQ sensor for 14 days. Glucose levels will be recorded.

SUMMARY:
This research project aims to investigate the everyday relevance of reactive hypoglycemia (hypoglycemia after a glucose load) in the oral glucose tolerance test (OGTT). Therefore, blood glucose profiles in everyday life will be examined using continuous glucose measurement (Free Style Libre PRO IQ system) over a period of 14 days in affected persons.

DETAILED DESCRIPTION:
The aim of this analysis is to examine people who underwent an OGTT due to various endocrinological and metabolic issues and developed reactive hypoglycemia, defined as a drop in blood glucose <70mg/dl during the course of the test. During OGTT routine laboratory testing will be performed as part of routine clinical practice. In order to investigate the occurrence and perception of hypoglycaemia in the everyday lives of those affected, their blood glucose profiles will be recorded and evaluated over a period of 14 days.

In addition, the perception of (suspected) hypoglycemia and counteraction will be documented. Anthropometric data will be recorded and a bioelectrical impedance analysis performed to check a correlation with the body composition. Subjects will be recruited via the endocrinology outpatient clinic as part of medical care. To date, very little CGM data are available on the frequency and extent of reactive hypoglycemia in the everyday lives of people without diabetes mellitus. Therefore, 20 subjects with hypoglycemia in the OGTT will be included in this exploratory pilot study for hypothesis generation in order to investigate the occurrence and perception of hypoglycemia in everyday life.

ELIGIBILITY:
Inclusion Criteria:

* hypoglycemia during a 75 g oral glucose tolerance test defined as glucose level below 70 mg/dl at timepoint 180 min.
* written consent

Exclusion Criteria:

* diabetes mellitus
* use of medication interfering with glucose metabolism (steroid, antidiabetic medications)
* surgery of upper GI-tract
* known plaster allergies
* any other clinical condition that would endanger participants safety or question scientific success according to the physicians opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of hypoglycemia | 14 days
  Occurrence of glucose levels below 70 mg/dl assessed by CGM.
Frequency of hypoglycemia | 14 days
  Number of glucose levels below 70 mg/dl assessed by CGM.
Severity of hypoglycemia | 14 days
  Non-severe hypoglycemia defined as glucose levels < 70 mg/dl but >= 54mg/dl; severe hypoglycemia defined as glucose levels < 54mg/dl assessed by CGM.

SECONDARY OUTCOMES:
Time of occurence of hypoglycemia | 14 days
  Occurence of hypoglycemia during day or night time and correspondence to food intake assessed by CGM.
Perception of hypoglycemia | 14 days
  Incidence of typical symptoms of hypoglycemia perceived by the participant, documented in a protocol with free-text fields handed out to the participant during 1st study visit.
Time in predefined glucose ranges | 14 days
  Time spent in the following glucose ranges: time above range: >140mg/dl; time in range: 71-140mg/dl; time below range: <70mg/dl; time with severe hypoglycemia: <54mg/dl assessed by CGM.
Mean glucose levels | 14 days
  Mean glucose levels during monitoring period assessed by CGM.
Glucose variability | 14 days
  Glucose variability during monitoring period assessed by CGM.
Correlation between severity of hypoglycemia during ogtt and hypoglycemia in everyday life | Varying time point between oGTT and 14 days of glucose assessment using CGM
  Correlation between severity of hypoglycemia during OGTT and incidence and severity of hypoglycemia in everyday life assessed by CGM.
Correlation between body composition and hypoglycemia in everyday life | 14 days
  Correlation between body composition (assessed by bioelectrical impedance analysis and anthropometric measurements) and incidence as well as severity of hypoglycemia in everyday life assessed by CGM.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, Prof., Principal Investigator — University Hospital Ulm
Locations (1):
- Universityhospital Ulm, Ulm, Germany